CLINICAL TRIAL: NCT01236911
Title: Prognosis Association of Hypocalcemia on Moderate-severe TBI, COHORTE STUDY
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Universidad Autonoma de San Luis Potosí (Other)
Responsible Party: Juan Manuel Viñas Rios, UASLP fACULTY OF MEDICINE
Other Study IDs: NCT071110
Record Dates: First submitted 2010-11-08; First posted 2010-11-09 (Estimated); Last update posted 2010-11-09 (Estimated); Status verified 2010-11

CONDITIONS: Calcium , Prognosis in Patients
Keywords: Calcium , TBI,complications, days in hospital

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Calcium after moderate-severe TBI: Patients with moderate -severe TBI with less as 24 hrs , admitted in emergency. We will measure seric calcium to compare the differences between both groups
  Interventions: Other: Calcium Measurement

INTERVENTIONS:
Other: Calcium Measurement — after moderate-severe TBI (less as 24 hrs)

SUMMARY:
Will have bad prognosis the patients with low calcium (less of 24 hrs of te admission in hospital)after moderate - severe TBI that the patients that do not developed this condition?

DETAILED DESCRIPTION:
Through the years the investigators have seen that the patients with low calcium after moderate-severe TBI had bad prognosis including more complications, and more days in hospital. The investigators want to make an association between the patients that developed this condition and the patients that do not developed this condition

ELIGIBILITY:
Inclusion Criteria:

* Man - woman between 16-65 years old with moderate -severe TBI less as 24 hrs,Count with tomographic study

Exclusion Criteria:

* Use of steroids, use of statins, Administration of Tromethamine, calcium antagonists, fibrates, niacin, cyclosporine, macrolides.
* Unclassifiable lesions in brainstem

Ages: 16 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients bettween 16 and 65 years old with moderate -severe TBI with less as 24 hours , without administration of steroids or statins
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2010-10; Primary Completion 2012-09 (Estimated); Study Completion 2012-11 (Estimated)

PRIMARY OUTCOMES:
Establishment an association between the patients that developed Hypocalcemia less 24 hrs after moderate-severe TBI with patients that did not develop this condition | 2 years

SECONDARY OUTCOMES:
Identify the more relevant prognosis factors | 2 years

CONTACTS AND LOCATIONS:
Locations (1):
- Juan Manuel Viñas Rios, San Luis Potosí City, San Luis Potosí, Mexico